CLINICAL TRIAL: NCT06228430
Title: A Single Dose, Randomized, Open-label, Two-way Crossover Bioequivalence Study of Generic Acyclovir 800 mg Tablet and Reference Product (ZoviraxTM) in Healthy Thai Volunteers Under Fasting Conditions
Brief Title: The Bioequivalence Study of Acyclovir 800 mg Tablet in Healthy Thai Volunteers Under Fasting Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Bio service (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: BE23-028
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteer
Keywords: Bioequivalence Study; Acyclovir
MeSH Terms: interventions — Acyclovir; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acyclovir 800 mg (Test Drug) (Experimental): Generic Acyclovir 800 mg Tablet
  Interventions: Drug: Acyclovir 800 mg Tablet; Drug: Zovirax™ 800 mg Tablet
- ZoviraxTM 800 mg Tablet (Reference Drug) (Active Comparator): ZoviraxTM 800 mg Tablet
  Interventions: Drug: Acyclovir 800 mg Tablet; Drug: Zovirax™ 800 mg Tablet

INTERVENTIONS:
Drug: Acyclovir 800 mg Tablet — Acyclovir 800 mg Tablet (Test Drug)
  Other Names: Acyclovir 800 mg
Drug: Zovirax™ 800 mg Tablet — Zovirax™ 800 mg Tablet (Reference Drug)
  Other Names: Acyclovir 800 mg

SUMMARY:
A Single Dose, Randomized, Open-label, Two-way Crossover Bioequivalence Study of Generic Acyclovir 800 mg Tablet and Reference Product (Zovirax™) in Healthy Thai Volunteers under Fasting Conditions

DETAILED DESCRIPTION:
This study is conducted to investigate bioequivalence information which is required to ensure therapeutic equivalence of a test product and a reference product as well as to be considered as one aspect of product quality. Bioequivalence is defined as the absence of a significant difference in the rate and extent to which the active ingredient or active moiety in pharmaceutical equivalents or pharmaceutical alternatives becomes available at the site of drug action when administered at the same molar dose under similar conditions in an appropriately designed study.

The manufacturer in Thailand needs to formulate a generic acyclovir 800 mg tablet. This study has been planned to evaluate the pharmacokinetics of this formulation and determine its bioequivalence with the reference product, Zovirax™, at the same dose.

ELIGIBILITY:
IInclusion Criteria

1. Healthy Thai male subjects between the ages of 18 to 55 years
2. Body mass index between 18.5 to 30.0 kg/m2
3. Normal laboratory values, including vital signs and physical examination, for all parameters in clinical laboratory tests at screening Any abnormalities from the normal or reference range will be carefully considered clinically relevant by the physician as individual cases, documented in study files prior to enrolling the subject in this study.
4. Male subjects who are willing or able to use effective contraceptive e.g. condom or abstinence after check-in in Period 1 until 7 days after the end of study in Period 2
5. Have voluntarily given written informed consent (signed and dated) by the subject prior to participating in this study

Exclusion Criteria

1. History of allergic reaction or hypersensitivity to alfuzosin or any of the other components of this product.
2. History or evidence of clinically significant renal, hepatic, gastrointestinal (e.g. intestinal occlusion), hematological, endocrine (e.g. hyper-/hypothyroid), pulmonary or respiratory (e.g. allergic rhinitis, asthma), cardiovascular (e.g. hyper-/hypotension), psychiatric (e.g. depression), neurologic (e.g. convulsant), allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) or any significant ongoing chronic medical illness.
3. Have high risk for coronavirus infection based on risk assessment questionnaire or diagnosed as confirmed case of COVID-19.
4. History about administration of COVID-19 vaccine within 30 days prior to check-in in each Period.
5. History or evidence of regular faintness, dizziness, headache or postural hypotension
6. History or evidence of galactose intolerance, the Lapp lactase deficiency or glucosegalactose malabsorption.
7. History of problems with swallowing tablet or capsule
8. History of sensitivity to heparin or heparin-induced thrombocytopenia.
9. Any condition possibly affecting drug absorption e.g. gastrectomy, enterectomy, gastritis or duodenal or gastric ulceration other than appendectomy
10. History of diarrhea or vomiting within 24 hours prior to check-in in each period
11. History or evidence of drug addict or investigation with urine sample shows a positive test for drug of abuse (morphine, marijuana or methamphetamine).
12. Have sitting systolic blood pressure of less than 90 mmHg or more than 139 mmHg and diastolic blood pressure of less than 60 mmHg or more than 89 mmHg on screening day and on the check-in day. If abnormal blood pressure detects, the measurement should be repeated two more times after take a rest for at least 5 minutes each. The last measurement value should be used to determine the subject's eligibility.
13. Investigation of vital signs shows pulse rate less than 60 or more than 100 beats per minute on screening day and on the check-in day. If abnormal pulse rate detects, the measurement should be repeated two more times after take a rest for at least 5 minutes each. The last measurement value should be used to determine the subject's eligibility
14. 12-lead ECG demonstrating QTc >450 msec, a QRS interval >120 msec or with an abnormality considered clinically significant at screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG will be repeated two more times and the average of the three QTc or QRS values will be used to determine the subject's eligibility
15. Investigation with blood sample shows positive test for HBsAg
16. Abnormal liver function, ≥1.5 times of upper normal limit of reference range for ALT, AST or bilirubin levels at screening laboratory test.
17. Have eGFR (CKD-EPI) < 30 mL/min/1.73 m2 based on serum creatinine results, at the screening laboratory test or during enrollment.
18. History or evidence of habitual use of tobacco or nicotine containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study.มีประวัติหรือหลักฐานของการสูบ
19. History or evidence of alcoholism or harmful use of alcohol (less than 2 years) i.e., alcohol consumption of more than 14 standard drinks per week for men (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 mL of 40% distilled spirits, such as rum, whisky, brandy, etc.).
20. History or evidence of alcohol consumption or alcohol-containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study or alcohol breath test shows positive result.In case of alcohol breath test result represents the alcohol concentration range of 1 - 10 mg% BAC and the physician carefully considers that the value came from other reasons, not from the alcohol drinking behavior of subjects, the test will be repeated two times separately, not more than 10 minutes. The result of the last time should be used for subject's eligibility which must be 0 mg%BAC.
21. History or evidence of habitual consume of tea, coffee, xanthine or caffeine containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study.
22. Consume or drink juice of grapefruit or orange or pomelo or its supplement / containing products and cannot abstain for at least 7 days prior to check-in in Period 1 and continued for entire duration of the study.
23. Use of prescription or nonprescription drugs (e.g. nitrates, paracetamol, erythromycin, clarithromycin, ketoconazole, itraconazole, prazosin, urapidil or minoxidil etc.), herbal medications or supplements (e.g. St. John's wort), vitamins or mineral (e.g. iron) or dietary supplements within 14 days prior to check-in in Period 1 and continued for entire duration of the study.
24. Participated in other clinical trials within 90 days prior to check-in in Period 1 (except for the subjects who drop out or withdrawn from the previous study prior to Period 1 dosing) or still participates in the clinical trial or participates in other clinical trials during enrollment in this study.
25. Blood donation or blood loss ≥ 1 unit (1 unit is equal to 350-450 mL of blood) within 90 days prior to check-in in Period 1 or during enrollment.
26. Subjects with poor venous access or intolerant to venipuncture
27. Unwilling or unable to comply with schedule visit, treatment plan and other study procedures until end of study.
28. Inability to communicate well (i.e. language problem, poor mental development, psychiatric illness or poor cerebral function) that may impair the ability to provide written informed consent or cooperate with clinical team.
29. Subjects who are employees of International Bio Service Co., Ltd., or Sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-12 (Estimated); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-22 (Estimated)

PRIMARY OUTCOMES:
Plasma Area Under the Curve (AUC(0 to 36 Hour)) for Acyclovir | Through 36 Hours Post Dose
  Plasma Area Under the Curve of Acyclovir
Peak Plasma Concentration (Cmax) of Acyclovir | 36 Hours Post Dose
  Peak Plasma Concentration (Cmax) for Acyclovir

CONTACTS AND LOCATIONS:
Overall Officials: Uthai Suvanakoot, Principal Investigator — International Bio service

IPD SHARING:
Plan to Share IPD: No